CLINICAL TRIAL: NCT03928977
Title: Contribution of Functional Imaging to the Diagnostic and Assesment of the Acute Phase of Transient Ischemic Attacks : a Preliminary Study
Brief Title: Functional Imaging in the Acute Phase of Transient Ischemic Attacks
Acronym: IMAGE AIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: P/2018/370
Record Dates: First submitted 2019-04-24; First posted 2019-04-26 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Transient Ischemic Attack
Keywords: Transient Ischemic Attack; Stroke; functional Magnetic Resonance Imaging
MeSH Terms: conditions — Ischemic Attack, Transient; Stroke | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Confirmed TIA (Other): Confirmed TIA at 3 months with standardized neurological expertise
  Interventions: Diagnostic Test: Functional Magnetic Resonance Imaging
- Confirmed non-TIA (Other): Not-confirmed TIA at 3 months with standardized neurological expertise
  Interventions: Diagnostic Test: Functional Magnetic Resonance Imaging

INTERVENTIONS:
Diagnostic Test: Functional Magnetic Resonance Imaging — fMRI sequences done with motor paradigm (right and left arm), followed by resting state acquisition

SUMMARY:
The aim of the study is to find a radiological biomarker of Transient Ischemic Attacks (TIA) thanks to functional Magnetic Resonance Imaging (fMRI) done within the 24 hour after symptoms onset.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted in for a transient neurologic deficit and suspicion of TIA of carotid circulation
* Prescription for conventionnal MRI

Exclusion Criteria:

* Contraindication to MRI
* Previous neurological disease (with lesions)
* Severe psychiatric disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-10-15 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Blood-Oxygen-Level Dependent signal | 24 hours after symptoms onset
  BOLD effect differences in motor cortex from pathological side versus healthy side measured by fMRI within the 24 hours after symptom onset, during a motor paradigm

SECONDARY OUTCOMES:
Resting state | 24 hours after symptoms onset
  Bold effect differences in resting state networks from pathological side versus healthy side measured by fMRI within the 24 hours after symptom onset, during a motor paradigm

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Besançon, Besançon, France